CLINICAL TRIAL: NCT00303342
Title: Neuroendocrine Mechanisms in Behavioral Treatment of Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sat Bir S. Khalsa, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AT002490 (NIH); R01AT002490 (NIH)
Record Dates: First submitted 2006-03-14; First posted 2006-03-16 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Insomnia
Keywords: sleep; arousal; stress; cortisol; catecholamines
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Desensitization, Psychologic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- mind body treatment (Experimental): regulation of attention, respiration and posture
  Interventions: Behavioral: mind body treatment
- desensitization (Active Comparator): mentation on insomnia behaviors and cognitive activity
  Interventions: Behavioral: desensitization

INTERVENTIONS:
Behavioral: mind body treatment — regulation of attention, respiration and posture
  Arms: mind body treatment
Behavioral: desensitization — mentation on insomnia behaviors and cognitive activity
  Arms: desensitization

SUMMARY:
The purpose of this study is to evaluate the change in measures of physiological arousal before and after behavioral treatment of insomnia.

DETAILED DESCRIPTION:
There is good evidence that physiological arousal, associated with sustained activation of the hypothalamic-pituitary axis and the sympathetic nervous system, is an underlying cause of chronic insomnia. Accordingly, relaxation-related treatments that address elevated cognitive and somatic arousal have been effective for insomnia. Previous studies have documented the effectiveness of behavioral treatments in reducing activation of the hypothalamic-pituitary axis and the sympathetic nervous system and in the treatment of specific medical disorders including insomnia. The aim of this proposal is to evaluate the hypothesis that improvements in chronic psychophysiological insomnia following a behavioral treatment are tightly associated with reduction of arousal in the hypothalamic-pituitary axis, as measured by plasma cortisol, and in the sympathetic nervous system, as measured by urinary catecholamines. Objective measures of sleep will be derived from polysomnographic recordings from subjects randomized into a 10-week active behavioral treatment or placebo behavioral control treatment group. Continuous 24-hour evaluation of cortisol and catecholamines will be performed under controlled laboratory conditions before and after treatment. We anticipate significant reductions in cortisol and catecholamines in the active treatment group as compared with the control group. We also anticipate that the active treatment will yield reductions in related measures of arousal including heart rate, autonomic arousal (as determined from heart rate variability), and body temperature. Given reported evidence that melatonin levels are chronically low in insomnia we anticipate an increase in the sleep-related hormone melatonin in the yoga treatment group. If achieved, these results will provide a novel demonstration of a reduction of arousal in a behavioral insomnia treatment and a behaviorally enhanced melatonin secretion under controlled laboratory conditions.

ELIGIBILITY:
Inclusion Criteria:

* primary insomnia for 6 months
* average total wake time >60 minutes and sleep efficiency <80%
* at least 1 daytime complaint due to insomnia
* adequate opportunity and circumstance for sleep

Exclusion Criteria:

* current psychiatric condition
* medical condition that interferes with sleep
* pregnancy
* rotating shift work, night work or transcontinental travel during study
* anticipated major life stressor over the course of the study
* use of hypnotic or psychoactive medications
* no idiopathic or sleep state misperception insomnia

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
plasma cortisol | pretreatment, posttreatment
plasma melatonin | pretreatment, posttreatment
urinary catecholamines | pretreatment, posttreatment
heart rate variability | pretreatment, posttreatment
subjective sleep efficiency | pretreatment, during treatment, posttreatment, followup
objective sleep efficiency | pretreatment, posttreatment

SECONDARY OUTCOMES:
actigraphy | pretreatment, posttreatment
EEG | pretreatment, posttreatment
subjective mood | pretreatment, during treatment, posttreatment, followup
depression | pretreatment, during treatment, posttreatment, followup
anxiety | pretreatment, during treatment, posttreatment, followup

CONTACTS AND LOCATIONS:
Overall Officials: Sat Bir S Khalsa, Ph.D., Principal Investigator — Brigham and Women's Hospital, Harvard Medical School
Locations (1):
- Sleep Disorders Program, Brigham and Women's Hospital, Boston, Massachusetts, United States